CLINICAL TRIAL: NCT06917911
Title: Phase II Study of Cytarabine + Daunorubicin (7 + 3) + Gemtuzumab Ozogamicin vs. Cytarabine + Daunorubicin (7 + 3) + Venetoclax for the Treatment of Newly Diagnosed Core Binding Factor Acute Myeloid Leukemia (CBF-AML) in Younger Adults: A MyeloMATCH Substudy
Brief Title: Testing the Addition of Venetoclax or Gemtuzumab Ozogamicin (GO) to Usual Treatment Regimen (Cytarabine and Daunorubicin, "7+3") for Core Binding Factor Acute Myeloid Leukemia (CBF-AML) to Improve Response (A MyeloMATCH Treatment Trial)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-02426; NCI-2025-02426 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MM1YA-A04 (Other: Alliance for Clinical Trials in Oncology); MM1YA-A04 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2025-04-08; First posted 2025-04-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Core Binding Factor Acute Myeloid Leukemia
MeSH Terms: interventions — Specimen Handling; Biopsy; Cytarabine; Daunorubicin; Gemtuzumab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regimen 1 (gemtuzumab ozogamicin 7+3) (Experimental): Patients receive gemtuzumab ozogamicin IV on days 1 and 4, cytarabine IV, continuously, on days 1-7 and daunorubicin IV on days 1-3 in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care consolidation/post-remission treatment at the discretion of the treating physician. Patients undergo echocardiography or MUGA scan during screening and bone marrow aspiration and biopsy and blood sample collection throughout the study. Patients may also undergo optional buccal swab collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Procedure: Echocardiography Test; Drug: Gemtuzumab Ozogamicin; Procedure: Multigated Acquisition Scan
- Regimen 2 (Venetoclax, 7+3) (Experimental): Patients receive venetoclax orally (PO) once daily (QD) on days 1-11, cytarabine IV, continuously, on days 2-8 and daunorubicin IV on days 2-4 in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care consolidation/post-remission treatment at the discretion of the treating physician. Patients undergo echocardiography or MUGA scan during screening and bone marrow aspiration and biopsy and blood sample collection throughout the study. Patients may also undergo optional buccal swab collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Drug: Venetoclax

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo optional buccal cell collection and/or blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
Drug: Gemtuzumab Ozogamicin — Given IV
  Other Names: Calicheamicin-Conjugated Humanized Anti-CD33 Monoclonal Antibody; CDP-771; CMA-676; gemtuzumab; hP67.6-Calicheamicin; Mylotarg; WAY-CMA-676
  Arms: Regimen 1 (gemtuzumab ozogamicin 7+3)
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto
  Arms: Regimen 2 (Venetoclax, 7+3)

SUMMARY:
This phase II MyeloMATCH treatment trial compares the effect of venetoclax to gemtuzumab ozogamicin, when given with cytarabine and daunorubicin ("7+3" regimen), for the treatment of patients with core binding factor acute myeloid leukemia (CBF-AML). Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Gemtuzumab ozogamicin is a monoclonal antibody, called gemtuzumab, linked to an antitumor antibiotic drug, called ozogamicin. Gemtuzumab is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of cancer cells, known as CD33 receptors, and delivers ozogamicin to kill them. Chemotherapy drugs, such as cytarabine and daunorubicin work in different ways to stop the growth of cancer cells either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving venetoclax with cytarabine and daunorubicin may have fewer side effects and be as effective or better than the combination with gemtuzumab ozogamicin in treating patients with core binding factor AML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Compare the rates of complete remission (CR) without measurable residual disease (CRMRD-) by multiparameter flow cytometry following induction therapy between the two treatment arms in each cohort separately.

SECONDARY OBJECTIVES:

I. To compare the rates of CR and composite complete remission (CRc) (CR+complete remission with incomplete hematologic recovery [CRi]+complete remission with partial hematologic recovery [CRh]) between the treatment arms.

II. To compare the overall survival (OS) between the treatment arms. III. To compare the event-free survival (EFS). IV. To compare cumulative incidence of relapse (CIR). V. To compare cumulative incidence of death (CID) between the treatment arms. VI. To compare the rate of early death at 30 days and 60 days between the treatment arms.

VII. To assess the rate and frequency of adverse events between treatment arms. VIII. To evaluate mutant RAS and mutant KIT as predictive biomarkers for CRMRD- rate in CBF AML.

EXPLORATORY OBJECTIVE:

I. To compare MRD (and its clinical implication, e.g., relapse rates) between flow cytometry (FC) and next generation sequencing (NGS)-based (RUNX1::RUNX1T1 or CBFB::MYH11).

CORRELATIVE OBJECTIVES:

I. To evaluate the frequency and clinical impact of variant allele frequency (VAF) of KIT mutation, KIT mutations in different exons (e.g., exon 8 or 17), CD33 expression, additional (secondary) mutations and cytogenetic abnormalities.

II. To evaluate the differences in clinical and molecular outcomes in patients with RUNX1::RUNX1T1 mutated versus CBFB::MYH11 mutated CBF AML.

OUTLINE: Patients are randomized to 1 of 2 regimens.

REGIMEN 1: Patients receive gemtuzumab ozogamicin intravenously (IV) on days 1 and 4, cytarabine IV, continuously, on days 1-7 and daunorubicin IV on days 1-3 in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care consolidation/post-remission treatment at the discretion of the treating physician. Patients undergo echocardiography or multigated acquisition (MUGA) scan during screening and bone marrow aspiration and biopsy and blood sample collection throughout the study. Patients may also undergo optional buccal swab collection throughout the study.

REGIMEN 2: Patients receive venetoclax orally (PO) once daily (QD) on days 1-11, cytarabine IV, continuously, on days 2-8 and daunorubicin IV on days 2-4 in the absence of disease progression or unacceptable toxicity. Patients then undergo standard of care consolidation/post-remission treatment at the discretion of the treating physician. Patients undergo echocardiography or MUGA scan during screening and bone marrow aspiration and biopsy and blood sample collection throughout the study. Patients may also undergo optional buccal swab collection throughout the study.

After completion of study treatment, patients are followed up at relapse and every 3 months for 2 years, then every 6 months until 5 years.

ELIGIBILITY:
Inclusion Criteria:

* GENERAL MYELOMATCH CRITERIA: Patients must be registered to the Master Screening and Reassessment Protocol and assigned to this protocol by the MATCHBox Treatment Verification Team
* GENERAL MYELOMATCH CRITERIA: Participants must not have received prior anti-cancer therapy for AML or myelodysplastic syndrome (MDS)

  * Note: Hydroxyurea to control the white blood cell count (WBC) and cytarabine up to 1 g/m^2 for urgent cytoreduction is allowed.
  * Note: Prior erythroid stimulating agent (ESA) is not considered prior therapy for the purposes of eligibility
* GENERAL MYELOMATCH CRITERIA: Participants must not receive any cytarabine-containing therapy other than up to 1 g/m^2 of cytarabine, which is allowed for urgent cytoreduction. The use of prior hydroxyurea, all-trans retinoic acid (ATRA), BCR-ABL directed tyrosine kinase inhibitor, erythropoiesis-stimulating agent, thrombopoietin receptor agonist and lenalidomide is allowed
* Diagnosis of AML with t(8;21)(q22;q22.1)/RUNX1::RUNX1T1 or AML with inv(16)(p13.1q22) or t(16;16)(p13.1;q22)/CBFB::MYH11. No FLT3 mutation (these patients should be considered for a FLT3-focused Myelomatch study)
* No prior AML or MDS-directed therapy except for urgent treatment of leukocytosis with leukapheresis, cytarabine, and hydroxyurea, Prior intrathecal chemotherapy for central nervous system (CNS) involvement of AML is permitted
* Age 18-59 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 3
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (unless patient has a history of Gilbert syndrome and direct bilirubin is ≤ 1.5 x ULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x upper limit of normal (ULN)
* Glomerular filtration rate (GFR) ≥ 30 mL/min/1.73m^2
* Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown. Therefore, for women of childbearing potential only, a negative urine or serum pregnancy test done ≤ 7 days prior to registration is required
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Participants with CNS disease are eligible for this trial and will be treated according to institutional guidelines with intrathecal chemotherapy for this aspect of their disease
* Patients with known HIV infection on effective anti-retroviral therapy with undetectable viral load within 6 months prior to registration are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* No known medical condition causing an inability to swallow oral formulations of agents

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Estimated)
Dates: Start 2026-02-18 (Estimated); Primary Completion 2027-11-25 (Estimated); Study Completion 2027-11-25 (Estimated)

PRIMARY OUTCOMES:
Complete remission without measurable residual disease (CRMRD-) | At end of induction (Up to 28 days)
  MRD will be evaluated by Molecular Diagnostics Network flow cytometry and will be defined at a threshold of < 10^-3.

SECONDARY OUTCOMES:
Rate of complete remission (CR) | At the end of treatment (Up to 28 days)
  Defined as the number of evaluable patients achieving a response of CR per European Leukemia Network (ELN) 2022 criteria at the end of treatment divided by the total number of evaluable patients. Rates of response will be compared between treatment arms using a chi-square test (or Fisher's exact test as needed). Point estimates will be generated for CR rate within each arm along with 95% confidence intervals using the Clopper-Pearson method.
Rate of composite CR | At the end of treatment (Up to 28 days)
  Defined as the number of evaluable patients achieving a response of CR or complete remission with incomplete hematologic recovery (CRi) or complete remission with partial hematologic recovery (CRh) per ELN 2022 criteria at the end of treatment divided by the total number of evaluable patients. Rates of response will be compared between treatment arms using a chi-square test (or Fisher's exact test as needed). Point estimates will be generated for CR rate within each arm along with 95% confidence intervals using the Clopper-Pearson method.
Overall survival (OS) | From registration until death due to any cause, up to 5 years
  The distribution of OS will be estimated using method of Kaplan-Meier. The median OS and 95% confidence interval will be reported.
Event free survival (EVS) | From randomization to induction failure, hematologic relapse from CR/CRh/CRi or death from any cause, whichever occurs first, up to 5 years
  Induction failure is defined as not achieving either CR, CRh or CRi by after induction therapy. The distribution of EFS will be estimated using method of Kaplan-Meier, and compared using log-rank tests. The median EFS and the corresponding 95% confidence interval will be reported.
Cumulative incidence of relapse (CIR) | From the date of achievement of a remission until the date of hematologic relapse, up to 5 years
  The distribution of CIR will be estimated using Fine-Gray model and reported via hazard ratios and 95% confidence interval with p values.
Cumulative incidence of death (CID) | From the date of achievement of a remission to death without prior relapse, up to 5 years
  The distribution of CID will be estimated using Fine-Gray model and reported via hazard ratios and 95% confidence interval with p values.
Rate of early death at 30 days (ED-30) | At 30 days
  ED-30 is defined as the total number of patients who died on or before day 30 from randomization divided by the total number of evaluable patients. Rate of early death at day 30 will be compared between treatment arms using a chi-square test (or Fisher's exact test as needed). Point estimates will be generated for ED-30 rate within each arm along with 95% confidence intervals using the Clopper-Pearson method.
Rate of early death at 60 days (ED-60) | At 60 days
  ED-60 is defined as the total number of patients who died on or before day 60 from randomization divided by the total number of evaluable patients. Rate of early death at day 60 will be compared between treatment arms using a chi-square test (or Fisher's exact test as needed). Point estimates will be generated for ED-60 rate within each arm along with 95% confidence intervals using the Clopper-Pearson method.
Incidence of adverse events | Up to 5 years
  As per national Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns. The incidence of severe (grade 3+) adverse events or toxicities will be described for each treatment arm and will also be compared between the arms. Fisher's exact tests will be used to quantitatively compare the incidence of severe as well as specific toxicities of interest between the treatment arms and we will graphically assess differences in maximum grades observed for toxicities between the arms.
Evaluate mutant RAS and mutant KIT as predictive biomarkers for CRMRD- rate | Up to 5 years
  In cohort 1, subgroup analysis will be conducted to evaluate the treatment effect among RAS mutated patients using Kaplan Meier methods and log-rank tests; similar subgroup analysis will be done among KIT mutated patients.

CONTACTS AND LOCATIONS:
Overall Officials: Celalettin Ustun, Principal Investigator — Alliance for Clinical Trials in Oncology

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm